CLINICAL TRIAL: NCT02292901
Title: Randomised Controlled Trial of Intubation With the McGrath Mac VideoLaryngoscope vs the Macintosh Laryngoscope
Brief Title: McGrath Mac VideoLaryngoscope vs the Macintosh Laryngoscope
Acronym: MGM-Eval
Status: Terminated | Phase: Not Applicable | Type: Interventional
Sponsor: Hopital Foch (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: 2013/42; 2013-A01307-38 (Other: ANSM)
Record Dates: First submitted 2014-11-12; First posted 2014-11-18 (Estimated); Last update posted 2016-10-31 (Estimated); Status verified 2016-10

CONDITIONS: Tracheal Intubation

STUDY DESIGN:
Who Masked: Participant
Oversight: Data Monitoring Committee: No

ARMS (2):
- Macintosh laryngoscope (Active Comparator): Tracheal intubation will be performed using a Macintosh laryngoscope
  Interventions: Device: Macintosh laryngoscope
- McGrath Mac videolaryngoscope (Experimental): Tracheal intubation will be performed using a McGrath Mac videolaryngoscope
  Interventions: Device: McGrath Mac videolaryngoscope

INTERVENTIONS:
Device: Macintosh laryngoscope
  Arms: Macintosh laryngoscope
Device: McGrath Mac videolaryngoscope
  Arms: McGrath Mac videolaryngoscope

SUMMARY:
Videolaryngoscopes become widely used. The aim of this study is to compare McGrath Mac videolaryngoscope to conventional MacIntosh laryngoscope in patients without known risk of difficult of mask ventilation and of tracheal intubation.

ELIGIBILITY:
Inclusion Criteria:

* patient scheduled for a general anesthesia with orotracheal intubation

Exclusion Criteria:

* predictable risk of difficult mask ventilation or of difficult tracheal intubation
* necessity of a rapid sequence induction
* contra-indication to sufentanil, to propofol, or to atracurium
* ENT, thoracic surgery, or intracranial surgery

Ages: 18 Years to 80 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 158 (Actual)
Dates: Start 2014-11; Primary Completion 2015-11 (Actual); Study Completion 2016-05 (Actual)

PRIMARY OUTCOMES:
Ease of tracheal intubation | 1 hour
  Ease of intubation is measured using the Intubation Difficulty Scale (Adnet et al. Anesthesiology 1997;87(6):1290-1297)

SECONDARY OUTCOMES:
Time to obtain the first capnogram (sec) | one hour
Score of Cormak and Lehane modified by Yentis | one hour
POGO (percentage of glottic opening) score | one hour
Rate of use of alternative techniques for intubation | one hour
Rate of esophageal intubation | one hour
Incidence of arterial oxygen desaturation (SpO2 <92%) | one hour
Rate of failure of tracheal intubation | one hour
Rate of hemodynamic abnormality | one hour
Postoperative throat pain | one day
Postoperative hoarseness | one day
Questionnaire of Salditt-Isabel | one hour

CONTACTS AND LOCATIONS:
Overall Officials: Michel Chandon, MD, Principal Investigator — Hopital Foch
Locations (2):
- France (2):
  - Institut Hospitalier Franco-Britannique, Levallois-Perret, Hauts de Seine
  - Hopital Foch, Suresnes, Hauts de Seine